CLINICAL TRIAL: NCT05737758
Title: An Assessment of Clinical Trial Experiences of Patients With Acne
Brief Title: Investigating Clinical Trial Participation for Acne Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 80343258
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Acne
Keywords: acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Participation in medical trials usually favors a particular demographic group. But there is limited research available to explain what trial attributes affect the completion of these specific demographic groups.

This trial will scrutinize the experiences of patients diagnosed with acne as they take part in a separate medical intervention clinical trial. The focus will be on tracking the rates of completion and withdrawal among these individuals.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future acne patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with acne
* Patient is able to read, understand and provide written Informed Consent
* Patient is a minimum of 18 years or older

Exclusion Criteria:

* Inability to perform regular electronic reporting
* Pregnant or lactating women
* Has significant intercurrent illness, psychiatric disposition or other factors that, in the opinion of the Investigator or Medical Monitor, precludes participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acne patients who are actively participating in a clinical study, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of acne patients who decide to join in a clinical study | 3 months
Rate of patients who remain in an acne clinical study to completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Eichenfield DZ, Sprague J, Eichenfield LF. Management of Acne Vulgaris: A Review. JAMA. 2021 Nov 23;326(20):2055-2067. doi: 10.1001/jama.2021.17633. PMID 34812859
- [Background] Williams HC, Dellavalle RP, Garner S. Acne vulgaris. Lancet. 2012 Jan 28;379(9813):361-72. doi: 10.1016/S0140-6736(11)60321-8. Epub 2011 Aug 29. PMID 21880356
- [Background] Titus S, Hodge J. Diagnosis and treatment of acne. Am Fam Physician. 2012 Oct 15;86(8):734-40. PMID 23062156

DOCUMENTS (1):
  • Informed Consent Form (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT05737758/ICF_000.pdf